CLINICAL TRIAL: NCT06769919
Title: A Randomized Controlled Study on the Efficacy and Safety of Neoadjuvant Radiotherapy Combined with Systemic Therapy for Early-stage Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WZ-1
Record Dates: First submitted 2025-01-03; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: radiotherapy; system therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: This study is a randomized, controlled, open-label clinical trial, planned to enroll 340 early-stage breast cancer patients with axillary lymph node biopsy-confirmed positivity. Participants will be divided into two groups. The control group will receive neoadjuvant systemic therapy, followed by surgery and adjuvant radiotherapy. The experimental group will receive neoadjuvant systemic therapy combined with neoadjuvant radiotherapy before undergoing surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adjuvant radiotherapy (No Intervention): receive neoadjuvant systemic therapy, followed by surgery and adjuvant radiotherapy
- Neoadjuvant radiotherapy (Experimental): receive neoadjuvant systemic therapy combined with neoadjuvant radiotherapy before undergoing surgery
  Interventions: Radiation: Neoadjuvant radiotherapy

INTERVENTIONS:
Radiation: Neoadjuvant radiotherapy — The experimental group will receive neoadjuvant systemic therapy combined with neoadjuvant radiotherapy before undergoing surgery
  Arms: Neoadjuvant radiotherapy

SUMMARY:
A total of 340 early-stage breast cancer patients with axillary lymph node biopsy-confirmed positivity were enrolled and divided into two groups. The control group received neoadjuvant systemic therapy followed by surgery and adjuvant radiotherapy. The experimental group received neoadjuvant systemic therapy and neoadjuvant radiotherapy followed by surgery. The treatment response of breast cancer, patient survival time, and treatment safety were subsequently evaluated.

DETAILED DESCRIPTION:
This study is a randomized, controlled, open-label clinical trial, planned to enroll 340 early-stage breast cancer patients with axillary lymph node biopsy-confirmed positivity. Participants will be divided into two groups. The control group will receive neoadjuvant systemic therapy, followed by surgery and adjuvant radiotherapy. The experimental group will receive neoadjuvant systemic therapy combined with neoadjuvant radiotherapy before undergoing surgery.

After providing full informed consent and signing the informed consent form, eligible participants will enter the trial period upon screening. Within 72 hours of enrollment confirmation, participants will begin neoadjuvant therapy. Patients in the control group will receive a neoadjuvant systemic therapy regimen selected by their physician, followed by surgery and adjuvant radiotherapy. Patients in the experimental group will receive both neoadjuvant systemic therapy and neoadjuvant radiotherapy. The radiotherapy regions will include the whole breast, supraclavicular and infraclavicular areas, and internal mammary regions, with a dose of 50 Gy over 25 fractions, plus a tumor bed boost of 10-16 Gy over 4-8 fractions.

Primary Endpoint:

Residual Cancer Burden (RCB) 0/I.

Secondary Endpoints:

Event-Free Survival (EFS) Invasive Disease-Free Survival (iDFS) Overall Survival (OS) Quality of life scores ECOG performance status scores Surgical incision healing scores Adverse Events (AEs)

Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for the trial:

1. Female patients aged ≥18 years and ≤65 years with newly diagnosed breast cancer;
2. Early-stage or locally advanced invasive breast cancer confirmed by histopathology according to the latest ASCO/CAP guidelines, meeting the following conditions:Axillary lymph node biopsy-positive;ECOG performance status score of 0-1;
3. Presence of at least one measurable lesion based on RECIST 1.1 criteria.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥18 years and ≤65 years；
* newly diagnosed breast cancer;
* Axillary lymph node biopsy-positive;
* ECOG performance status score of 0-1;

Exclusion Criteria:

* metastatic breast cancer or bilateral breast cancer;
* inflammatory breast cancer;
* Pregnancy and Lactation;

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Residual Cancer Burden (RCB) 0/I | From enrollment to the end of treatment at 8 weeks
  Residual Cancer Burden (RCB) is a standardized method used to quantify the amount of residual disease in breast cancer patients after neoadjuvant therapy (treatment given before surgery). It is calculated based on the size of the primary tumor, the cellularity of the tumor bed, and the extent of lymph node involvement. RCB is divided into four categories:
  RCB-0: Pathologic complete response (pCR), meaning no residual invasive cancer is found in the breast or lymph nodes.
  RCB-I: Minimal residual disease, indicating a very small amount of cancer remains after treatment.
  RCB-II: Moderate residual disease. RCB-III: Extensive residual disease. RCB-0 and RCB-I are often associated with better prognoses and higher survival rates compared to RCB-II and RCB-III

SECONDARY OUTCOMES:
Event-Free Survival (EFS) | From enrollment to 10 years later or death.
  Event-Free Survival (EFS) is defined as the time from randomization to the occurrence of any event, including disease progression, discontinuation of treatment for any reason, or death.
Invasive Disease-Free Survival (iDFS) | From enrollment to 10 years later or death.
Overall Survival (OS) | From enrollment to 10 years later or death.
Quality of life scores | From enrollment to 3 years after treatment completion.
ECOG performance status scores | From enrollment to 3 years after treatment completion.
Surgical incision healing scores | From enrollment to 1 years after treatment completion.
Adverse Events (AEs) | From enrollment to 3 years after treatment completion.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided